CLINICAL TRIAL: NCT01283074
Title: Prognostic Factors of Long-term Response to Treatment With Pegylated Interferon Alfa-2a in Patients With HbeAg-negative Chronic Hepatitis B. (Perseas)
Brief Title: An Observational Study of Pegasys (Peginterferon Alfa-2a) in Patients With HbeAg-negative Chronic Hepatitis B (Perseas)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22016
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational, multi-center, open-label study will evaluate the prognostic factors of long-term-response and the safety of Pegasys (peginterferon alfa-2a) in patients with HbeAg-negative chronic hepatitis B. Data will be collected for 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Diagnosis of HBeAg-negative chronic hepatitis B with compensated hepatic disease, virus multiplication, raised alanine amino transferase results and/or fibrosis

Exclusion Criteria:

* Co-infection with hepatitis A, C or D
* Co-infection with human immunodeficiency virus (HIV)
* Severe hepatic dysfunction or decompensated liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B on treatment with Pegasys
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2009-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with combined (virological and biochemical) response | 48 weeks after end of treatment

SECONDARY OUTCOMES:
Normalization of serum alanine aminotransferase | 12 months
Safety (Incidence of adverse events) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Greece (7):
  - Alexandroupoli
  - Athens
  - Larissa
  - Pátrai
  - Piraeus
  - Rhodes
  - Thessaloniki

REFERENCES:
- [Derived] Goulis I, Karatapanis S, Akriviadis E, Deutsch M, Dalekos GN, Raptopoulou-Gigi M, Mimidis K, Germanidis G, Drakoulis C, Triantos C, Zintzaras E, Bakalos G, Papatheodoridis G. On-treatment prediction of sustained response to peginterferon alfa-2a for HBeAg-negative chronic hepatitis B patients. Liver Int. 2015 May;35(5):1540-8. doi: 10.1111/liv.12725. Epub 2014 Nov 20. PMID 25368957